CLINICAL TRIAL: NCT02404883
Title: Decisional Conflict of Young Cancer Patients With Regard to Fertility Preservation - Effects of an Online Decision-aid Tool
Brief Title: Decisional Conflict of Young Cancer Patients With Regard to Fertility Preservation
Acronym: Fertionco
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss Bridge (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-265
Record Dates: First submitted 2015-03-19; First posted 2015-04-01 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Cancer
Keywords: Cancer; decisional conflict; online; decision-aid tool
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): care as usual (fertility preservation counseling)
- intervention group (Experimental): Intervention: use of an online decision-aid tool after fertility preservation counseling
  Interventions: Other: Online Decision-Aid Tool

INTERVENTIONS:
Other: Online Decision-Aid Tool
  Arms: intervention group

SUMMARY:
Women who are diagnosed with cancer during their reproductive lifespan might be confronted with impaired fertility. Nowadays a number of fertility preservation options are available. Decisions about whether and how to protect fertility have to be made in a very short time period, right after cancer diagnosis and before start of treatment. The psychological impact for patients is considerable. This project aims at developing a standardized decision-aid tool to support the decision-making process about fertility preservation in young cancer patients. It is designed as an online decision-aid tool. A web-based tool is perfectly designed for this target group and offers new possibilities providing flexible and individually tailored information.

The aim of the study is to examine the benefits of the online decision-aid tool compared with standard counseling (usual care). Decisional conflict is measured immediately after counseling as well as one month later. One year after counseling, decisional regret is being evaluated additionally. If the decision-aid tool proves to be helpful and useful, the online design allows making it available for a wide range of concerned patients.

DETAILED DESCRIPTION:
Background: Impaired fertility is often a consequence of successful cancer treatment and fertility preservation (FP) is nowadays an option for young cancer survivors. Decisions on FP, however, have to be made in the short time period after cancer diagnosis and before onset of treatment. According to previous studies the availability of helpful information is still low, decisional conflict substantial and decisions-aids would be highly desirable.

Objectives: The project aims at introducing the knowledge gained by the previous research into the development of a standardized online decision aid (DA) that complements and supports shared decision-making in fertility issues and FP for young cancer patients and their medical caretakers and to evaluate the efficacy of this DA compared with usual care. Primary objective: To show that an online decision-aid tool in addition to standard counselling reduces decisional conflict compared to standard counselling alone. Secondary objectives: 1) to assess whether the decision-aid tool decreases decisional regret significantly, 2) to assess whether the use of the decision-aid tool increases the patients' knowledge on FP and 3) to assess whether patients estimate the decision-aid tool helpful in facilitating the decision-making process.

Methods: Design: Prospective, consecutive interventional study comparing a control group with standard counselling (phase 1) with an interventional group with counselling and application of the DA (phase 2). After completing phase 1 and 2 with a sample of 40 participants, we change the study design into a randomized controlled trial and randomize 88 participants in this part of the study. Sample: A total of 120 young cancer patients followed at one of the collaborating Swiss or German cancer centers aged 16 to 40 years who are possible candidates for FP . Intervention: Online DA, which is developed based on the applicants' research findings and on a prospectively evaluated fertility-related Australian decision aid booklet. Measures: Decisional Conflict Scale (DCS); items on knowledge, attitude and willingness concerning FP; decision regret scale (DRS); items on satisfaction and helpfulness of the DA.

Procedures: The control and the interventions group completes the questionnaires at three time points, i.e. immediately after the counselling (T1), after 1 month (T2) and after 12 months (T3).

Analysis and statistics: The difference in decisional conflict between the two groups will be analyzed by using a one-way analysis of variance (ANOVA) and a propensity score weighted ANOVA to adjust for confounding variables.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Age 16 to 40 years
* German speaking
* Access to a computer
* Pre-menopausal at time of diagnosis
* Not yet having started (adjuvant) cancer therapy
* family planning not completed

Exclusion Criteria:

- Cancer treatment not affecting reproductive function

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 79 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
change (reduction) of decisional conflict (Decisional Conflict Scale) | 3 times: within 5 days after fertility preservation counseling, one month after counseling, 12 month after counseling
  with the

SECONDARY OUTCOMES:
change (reduction) of decisional regret (Decisional Regret Scale) | twice: 1 month after fertility preservation counseling, 12 month after counseling
  with the Decisional Regret Scale
change (increase) of knowledge about fertility preservation (questionnaire) | twice: within 5 days after fertility preservation counseling, 1 month after counseling
  with a questionnaire which assess the knowledge about various fertility preservation methods
helpfulness and satisfaction of decision-aid tool (questionnaire) | twice: within 5 days after fertility preservation counseling, 1 month after counseling
  questionnaire to assess helpfulness and satisfaction of tool only for the intervention group, who used the decision-aid tool

CONTACTS AND LOCATIONS:
Overall Officials: Sibil Tschudin, PD Dr. med., Principal Investigator — Universitätsspital Basel Frauenklinik
Locations (1):
- Universitätsspital Frauenklinik, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Ehrbar V, Urech C, Rochlitz C, Zanetti Dallenbach R, Moffat R, Stiller R, Germeyer A, Nawroth F, Dangel A, Findeklee S, Tschudin S. Randomized controlled trial on the effect of an online decision aid for young female cancer patients regarding fertility preservation. Hum Reprod. 2019 Sep 29;34(9):1726-1734. doi: 10.1093/humrep/dez136. PMID 31398258